CLINICAL TRIAL: NCT00707980
Title: A Long-Term, Open-Label, Flexible-Dose, Extension Study Evaluating the Safety and Tolerability of Lu AA21004 in Subjects With Major Depressive Disorder
Brief Title: Safety and Tolerability of Vortioxetine (Lu AA21004) in Adults With Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LuAA21004_301; 2008-001581-91 (EudraCT Number); U1111-1113-9564 (Registry Identifier: WHO)
Record Dates: First submitted 2008-06-27; First posted 2008-07-02 (Estimated); Results first posted 2013-12-13 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-10

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Depression; Melancholia; Mood Disorder; Dysthymic Disorder; Drug Therapy
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Depressive Disorder; Mood Disorders; Dysthymic Disorder | interventions — Vortioxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vortioxetine (Experimental): Vortioxetine 2.5 mg, 5 mg or 10 mg, encapsulated tablets, orally, once daily for up to 52 weeks. For the first week of treatment all participants received 5 mg/day vortioxetine, thereafter, the dose could be increased to 10 mg/day or decreased to 2.5 mg/day, based on participant's response and tolerability as judged by the investigator.
  Interventions: Drug: Vortioxetine

INTERVENTIONS:
Drug: Vortioxetine — Encapsulated vortioxetine immediate-release tablets
  Other Names: Lu AA21004; Brintellix®

SUMMARY:
The purpose of this study is to determine the long-term efficacy and safety of vortioxetine, once daily (QD), in adults with major depressive disorder.

DETAILED DESCRIPTION:
The drug that was tested in this study is called vortioxetine. Vortioxetine is being tested to treat depression in people who have major depressive disorder (MDD). This study looked at MDD relief in people who took vortioxetine.

The study enrolled 836 patients that had completed one of two other vortioxetine studies. Participants received 5 mg of vortioxetine for the first week of treatment. After completing the first week of treatment, the dose could be increased to 10 mg/day or decreased to 2.5 mg/day based on participant's response as judged by the doctor.

All participants were asked to take one encapsulated tablet at the same time each day throughout the study.

This multi-center trial was conducted worldwide. The overall time to participate in this study was up to 56 weeks. Participants made 13 visits to the clinic, and were contacted by telephone 4 weeks after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Has completed the double blind treatment period of either study Lu AA21004_304 (NCT00672620) or LuAA21004_305 (NCT00735709) immediately prior to enrollment in the extension study (ie, the baseline visit is the same visit as the completion visit of the double blind treatment of the preceding protocol).
* Suffers from a major depressive episode as the primary diagnosis according to Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR) criteria (classification code 296.xx) at entry into the prior Lu AA21004_304 or Lu AA21004_305 study.

Exclusion Criteria:

* In addition to meeting the exclusion criteria for studies Lu AA21004_304 or Lu AA21004_305 at the time of enrollment into those studies respectively, with the exception of the criteria prohibiting previous exposure to Lu AA21004 and investigational drugs, and the criteria prohibiting patients with increased intraocular pressure, or risk of acute narrow-angle glaucoma, the following exclusion criteria apply:

  * Has Major Depressive Disorder for whom other psychiatric disorders (mania, bipolar disorder, schizophrenia, or any psychotic disorder) have been diagnosed during the prior study.
  * The participant, in the investigator's opinion, has a significant risk of suicide and/or a score of ≥5 points on item 10 (suicidal thoughts) of the Montgomery Åsberg Depression Rating Scale.
  * The participant, in the opinion of the investigator, is unlikely to comply with the clinical study protocol or is unsuitable for any reason.
  * Has a clinically significant moderate or severe ongoing adverse event related to study medication from the prior study.
  * Has used/uses disallowed concomitant medication.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 836 (Actual)
Dates: Start 2008-06; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Clinical Science, Study Director — Takeda
Locations (92):
- United States (38):
  - Beverly Hills, California
  - Irvine, California
  - Santa Ana, California
  - Torrance, California
  - Upland, California
  - Bradenton, Florida
  - Coral Springs, Florida
  - Fort Walton Beach, Florida
  - Gainesville, Florida
  - Jacksonville, Florida
  - Maitland, Florida
  - Orlando, Florida
  - South Miami, Florida
  - West Palm Beach, Florida
  - Atlanta, Georgia
  - Smyrna, Georgia
  - Chicago, Illinois
  - Libertyville, Illinois
  - Oak Brook, Illinois
  - Prairie Village, Kansas
  - Owensboro, Kentucky
  - Baltimore, Maryland
  - Pittsfield, Massachusetts
  - Worcester, Massachusetts
  - Flowood, Mississippi
  - New York, New York
  - Olean, New York
  - Beachwood, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Allenport, Pennsylvania
  - Lancaster, Pennsylvania
  - Memphis, Tennessee
  - Austin, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Seattle, Washington
  - Milwaukee, Wisconsin
- Australia (3):
  - Elizabeth Vale
  - Richmond
  - Southport
- Croatia (2):
  - Osijek
  - Zagreb
- France (3):
  - Bully-les-Mines
  - Marseille
  - Strasbourg
- Germany (8):
  - Berlin
  - Bochum
  - Chemnitz
  - Hüttenberg
  - Leipzig
  - München
  - Nuremberg
  - Wiesbaden
- Latvia (3):
  - Liepāja
  - Riga
  - Sigulda
- Lithuania (2):
  - Šiauliai
  - Vilnius
- Kuala Lumpur, Malaysia
- Netherlands (3):
  - SchHoogfliet
  - Wildervank
  - Zwijndrecht
- Poland (6):
  - Bialystok
  - Leszno
  - Pruszków
  - Skórzewo
  - Torun
  - Tuszyn
- Russia (7):
  - Moscow
  - Nizhny Novgorod
  - Novosibirsk
  - Omsk
  - Saint Petersburg
  - Stavropol
  - Tomsk
- Belgrade, Serbia
- South Africa (5):
  - Bryanston
  - Durban
  - Lyttelton
  - Noordheuwel
  - Pretoria
- South Korea (4):
  - Buchon
  - Gyeonggi-do
  - Incheon
  - Seoul
- Kaohsiung City, Taiwan
- Ukraine (4):
  - Dnipro
  - Kiev
  - Luhansk
  - Simferopol
- Glasgow, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 88 investigative sites in Australia, Croatia, France, Germany, Korea, Latvia, Lithuania, Malaysia, The Netherlands, Poland, Russia, Taiwan, Ukraine, and the United States from 17 June 2008 to 23 August 2010.
Pre-assignment Details: Participants who completed short-term efficacy and safety studies Lu AA21004_304 (NCT00672620) and LuAA21004_305 (NCT00735709) were eligible to receive the 52-week treatment with vortioxetine in this open-label extension study.
Period: Overall Study
Arm/Group | Vortioxetine
Started | 836
Received Treatment | 834
Completed | 526
Not Completed | 310
Not completed — Adverse Event | 49
Not completed — Lack of Efficacy | 35
Not completed — Non-Compliance with Study Drug | 28
Not completed — Protocol Deviations | 19
Not completed — Withdrawal of Consent | 81
Not completed — Lost to Follow-up | 59
Not completed — Other | 39

BASELINE CHARACTERISTICS:
Arm/Group | Vortioxetine
Number analyzed (Participants) | 836
Age Continuous [Mean (Standard Deviation); unit: Years] | 45.5 (12.78)
Age, Customized [Number; unit: Participants]
  ≤55 years | 636
  >55 years | 200
Sex: Female, Male [Count of Participants; unit: Participants] — Note: Baseline refers to the open-label extension study baseline throughout these results.
  Participants
    Female | 526
    Male | 310
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian (White, including Hispanic) | 693
  Black | 86
  Asian | 54
  American Indian or Alaska Native | 2
  Native Hawaiian/ Other Pacific Islander | 1
Race/Ethnicity, Customized [Number; unit: Participants] — Race data available for 836 participants.
  Participants
    Hispanic/Latino | 53
    Non-Hispanic/Non-Latino | 782
    Missing | 1
Region of Enrollment [Number; unit: Participants]
  Australia | 4
  Germany | 207
  France | 11
  Croatia | 11
  Republic of Korea | 25
  Lithuania | 10
  Latvia | 20
  Malaysia | 17
  Netherlands | 7
  Poland | 57
  Russia | 40
  Taiwan | 3
  Ukraine | 37
  United States | 387
Weight [Mean (Standard Deviation); unit: kg] | 81.16 (20.829)
Height [Mean (Standard Deviation); unit: cm] | 169.00 (9.777)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.41 (7.074)
24-item Hamilton Depression Scale total score [Mean (Standard Deviation); unit: scores on a scale] — The 24-item Hamilton Depression Scale (HAM-D24) is a clinician-rated 24-item scale for assessing the severity of depression symptoms. The scores for each item range from 0 to 4 or 0 to 2, where 0 represents no symptoms. The rating is based on the past 7 days prior to the time of assessment. The total score ranges from 0 to 74, where a higher score indicates a greater depressive state.
  scores on a scale | 17.6 (9.40)
Montgomery Åsberg Depression Rating Scale (MADRS) total score [Mean (Standard Deviation); unit: scores on a scale] — The Montgomery Åsberg Depression Rating Scale (MADRS) is a depression rating scale consisting of 10 items, each rated 0 to 6. The 10 items represent the core symptoms of depressive illness. The overall score ranges from 0 (symptoms absent) to 60 (severe depression).
  scores on a scale | 16.6 (9.24)
Hamilton Anxiety Scale total score [Mean (Standard Deviation); unit: scores on a scale] — Hamilton Anxiety Scale (HAM-A) is an anxiety rating scale consisting of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behavior at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total scores range from 0 to 56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe. Total scores above 30 are rare, but indicate very severe anxiety.
  scores on a scale | 12.1 (7.17)
Clinical Global Impression - Severity scale score [Mean (Standard Deviation); unit: scores on a scale] — The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale where the clinician rates the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis on the following scale: 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
  scores on a scale | 3.2 (1.26)

OUTCOME MEASURES:

1. Primary Outcome: Physical Examination Findings
Description: Physical examination consisted of the following body systems: (1) appearance; (2) extremities; (3) skin; (4) head and neck; (5) eyes, ears, nose, and throat; (6) lungs and chest; (7) heart and cardiovascular system; (8) abdomen; and (9) musculoskeletal system. An assessment of the nervous system was conducted; any findings were captured under the appropriate body area.
  Each system was assessed as normal or abnormal.
Time Frame: Baseline and Week 52
Population: The safety set included all participants who enrolled and received at least 1 dose of open-label study medication. Results include data for participants with available data at each time point; 834 participants at Baseline and 524 participants at Week 52.
Measure: Number; unit: participants
Arm/Group | Vortioxetine
Number analyzed (Participants) | 834
participants
  Appearance at Baseline: Normal | 758
  Appearance at Baseline: Abnormal | 76
  Appearance at Week 52: Normal | 484
  Appearance at Week 52: Abnormal | 40
  Extremities at Baseline: Normal | 806
  Extremities at Baseline: Abnormal | 28
  Extremities at Week 52: Normal | 511
  Extremities at Week 52: Abnormal | 13
  Skin at Baseline: Normal | 730
  Skin at Baseline: Abnormal | 104
  Skin at Week 52: Normal | 465
  Skin at Week 52: Abnormal | 59
  Head-Neck at Baseline: Normal | 822
  Head-Neck at Baseline: Abnormal | 12
  Head-Neck at Week 52: Normal | 518
  Head-Neck at Week 52: Abnormal | 6
  Eyes-Ears-Nose-Throat at Baseline: Normal | 772
  Eyes-Ears-Nose-Throat at Baseline: Abnormal | 62
  Eyes-Ears-Nose-Throat at Week 52: Normal | 485
  Eyes-Ears-Nose-Throat at Week 52: Abnormal | 39
  Lungs-Chest at Baseline: Normal | 827
  Lungs-Chest at Baseline: Abnormal | 7
  Lungs-Chest at Week 52: Normal | 523
  Lungs-Chest at Week 52: Abnormal | 1
  Heart/Cardiovascular at Baseline: Normal | 816
  Heart/Cardiovascular at Baseline: Abnormal | 18
  Heart/Cardiovascular at Week 52: Normal | 512
  Heart/Cardiovascular at Week 52: Abnormal | 12
  Abdomen at Baseline: Normal | 818
  Abdomen at Baseline: Abnormal | 12
  Abdomen at Baseline: Not done | 4
  Abdomen at Week 52: Normal | 515
  Abdomen at Week 52: Abnormal | 8
  Abdomen at Week 52: Not done | 1
  Musculoskeletal at Baseline: Normal | 790
  Musculoskeletal at Baseline: Abnormal | 44
  Musculoskeletal at Week 52: Normal | 493
  Musculoskeletal at Week 52: Abnormal | 31

2. Primary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Evaluation Findings
Description: Participants with at least one post-baseline potentially clinically significant (as defined in the table below) serum chemistry, hematology or urinalysis result. ULN = upper limit of normal; LLN = Lower limit of normal.
Time Frame: Weeks 4, 8, 12, 20, 28, 36, 44 and 52
Population: Safety set
Measure: Number; unit: participants
Arm/Group | Vortioxetine
Number analyzed (Participants) | 834
participants
  Alanine aminotransferase (ALT) ≥ 3 X ULN | 3
  Aspartate aminotransferase (AST) ≥ 3 X ULN | 6
  Bilirubin ≥ 34.2 μmol/L | 1
  Cholesterol ≥ 7.8 mmol/L | 49
  Creatine kinase ≥ 2 X ULN | 80
  Creatinine ≥ 175 μmol/L | 1
  Glucose ≤ 2.8 mmol/L | 9
  Glucose ≥ 13.9 mmol/L | 7
  High density lipoprotein cholesterol < 0.9 mmol/L | 102
  Low density lipoprotein cholesterol ≥ 5.0 mmol/L | 69
  Potassium ≤ 3.0 mmol/L | 0
  Potassium ≥ 5.5 mmol/L | 45
  Sodium ≤ 125 mmol/L | 1
  Sodium ≥ 155 mmol/L | 1
  Triglycerides ≥ 3.40 mmol/L | 168
  Urate ≤ 0.7 X LLN | 4
  Urate ≥ 1.3 XULN | 12
  Eosinophils ≥ 0.6 10^9/L | 24
  Erythrocytes ≤ 0.9 X LLN | 9
  Erythrocytes ≥ 1.1 X ULN | 1
  Hematocrit ≤ 0.9 X LLN | 16
  Hemoglobin ≤ 0.9 X LLN | 41
  Leukocytes ≤ 2.8 X 10^9/L | 10
  Leukocytes ≥ 16 X 10^9/L | 3
  Lymphocytes ≤ 0.6 X 10^9/L | 5
  Lymphocytes ≥ 7 X 10^9/L | 0
  Neutrophils ≤ 1.4 X 10^9/L | 26
  Neutrophils ≥ 15 X 10^9/L | 2

3. Primary Outcome: Number of Participants With Potentially Clinically Significant Electrocardiogram (ECG) Findings
Description: A standard 12-lead ECG was performed at the designated study visits. The central reader reviewed and recorded the intervals (PR, QRS, RR, QT, and corrected QT interval [QTc]), and interpreted the ECG using 1 of the following categories: within normal limits or abnormal. The number of participants with at least one post-baseline potentially clinically significant ECG finding is reported. bpm = beats per minute; QTcB = QT interval corrected using Bazett's formula; QTcF = QT interval corrected using Fridericia's formula.
Time Frame: Weeks 4, 12, 24, 36 and 52
Population: Safety set
Measure: Number; unit: participants
Arm/Group | Vortioxetine
Number analyzed (Participants) | 834
participants
  Heart rate ≤50 bpm and change ≤-15bpm | 9
  Heart rate ≥120 bpm and change ≥15 bpm | 0
  RR interval <500 msec and change ≤-200 msec | 0
  RR interval >1200 msec and change ≥200 msec | 13
  PR interval <120 msec | 31
  PR interval ≥250 msec | 2
  QT interval <280 msec | 0
  QT interval >500 msec | 2
  QTcB <340 msec | 0
  QTcB >500 msec | 3
  QTcB Change <-60 msec | 6
  QTcB Change >60 msec | 4
  QTcF <340 msec | 0
  QTcF >500 msec | 2
  QTcF Change <-60 msec | 3
  QTcF Change >60 msec | 2

4. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: The intensity (severity) of each AE was defined as:
  * Mild: caused minimal discomfort and did not interfere in a significant manner with normal activities.
  * Moderate: sufficiently uncomfortable to produce some impairment of normal activities.
  * Severe: incapacitating, preventing the patient from participating in normal activities.
  The causal relationship between an AE and study drug was assessed by the investigator as Probable, Possible or Not Related; Related=AEs with causality of Possibly or Probably. A serious AE (SAE) was defined as any untoward medical occurrence that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, led to a congenital anomaly/birth defect, or was an important medical event that either jeopardized the patient, required intervention to prevent any of the SAEs defined above, a suicide attempt or an abortion.
Time Frame: From the first dose of open-label study drug until 4 weeks after the last dose (up to 56 weeks)
Population: Safety set
Measure: Number; unit: participants
Arm/Group | Vortioxetine
Number analyzed (Participants) | 834
participants
  Any adverse event | 589
  Related adverse event | 413
  Not related adverse event | 176
  Mild adverse event | 187
  Moderate adverse event | 320
  Severe adverse event | 82
  Adverse event leading to early termination | 50
  Serious adverse event | 29
  Serious related adverse event | 5
  Serious not related adverse event | 33
  Serious adverse event leading to early termination | 11
  Deaths | 0

5. Primary Outcome: Number of Participants With Potentially Clinically Significant Vital Sign Findings
Description: Participants with at least one potentially clinically significant post-baseline vital sign finding. The definition of clinically significant is included in the table below for each parameter. SSBP = supine systolic blood pressure; SDBP = supine diastolic blood pressure.
Time Frame: Weeks 1, 2, 4, 8, 12, 16, 20, 24, 28, 36, 44 and 52
Population: Safety set
Measure: Number; unit: participants
Arm/Group | Vortioxetine
Number analyzed (Participants) | 834
participants
  SSBP ≤90 mmHg and decrease of ≥20 mmHg | 7
  SSBP ≥180 mmHg and increase of ≥20 mmHg | 4
  SDBP ≤50 mmHg and decrease of ≥15 mmHg | 1
  SDBP ≥105 mmHg and increase of ≥15 mmHg | 8
  Supine pulse rate ≤50 bpm and decrease of ≥15 bpm | 7
  Supine pulse rate ≥120 bpm and increase of ≥15 bpm | 2
  Weight Change of ≥7% weight | 155

6. Secondary Outcome: Change From Baseline in Hamilton Depression Scale-24 Item (HAM-D24) Total Score
Description: The HAM-D24 is a clinician-rated 24-item scale for assessing the severity of depression symptoms. The scores for each item range from 0 to 4 or 0 to 2, where 0 represents no symptoms. The rating is based on the past 7 days prior to the time of assessment. The total score ranges from 0 to 74 where a higher score indicates a greater depressive state. Final Visit includes data from Week 52 or earlier for participants who didn't complete the 52 weeks.
Time Frame: Baseline and Weeks 1, 2, 4, 8, 12, 16, 20, 24, 28, 36, 44 and 52.
Population: Participants in the safety analysis set who had at least 1 post-baseline efficacy measurement, and with available data. "n" indicates the number of patients included in the analysis at each time point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Vortioxetine
Number analyzed (Participants) | 829
scores on a scale
  Week 1 (n=805) | -1.1 (5.27)
  Week 2 (n=822) | -3.1 (6.10)
  Week 4 (n=805) | -4.7 (7.07)
  Week 8 (n=752) | -6.5 (7.43)
  Week 12 (n=715) | -7.0 (8.27)
  Week 16 (n=671) | -7.7 (8.45)
  Week 20 (n=639) | -8.4 (8.51)
  Week 24 (n=613) | -8.3 (8.92)
  Week 28 (n=599) | -8.9 (8.91)
  Week 36 (n=568) | -9.3 (9.05)
  Week 44 (n=540) | -9.6 (9.32)
  Week 52 (n=522) | -10.0 (8.86)
  Final Visit (n=829) | -7.9 (9.66)

7. Secondary Outcome: Change From Baseline in the Montgomery Åsberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS is a depression rating scale consisting of 10 items, each rated 0 to 6. The 10 items represent the core symptoms of depressive illness. The overall score ranges from 0 (symptoms absent) to 60 (severe depression). Decrease in the total score or on individual items indicates improvement. Final Visit includes data from Week 52 or earlier for participants who didn't complete the 52 weeks.
Time Frame: Baseline and Weeks 4, 24 and 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Vortioxetine
Number analyzed (Participants) | 818
scores on a scale
  Week 4 (n=818) | -4.5 (7.38)
  Week 24 (n=642) | -7.9 (9.24)
  Week 52 (n=526) | -9.5 (8.90)
  Final Visit (n=818) | -7.4 (9.81)

8. Secondary Outcome: Change From Baseline in the Hamilton Anxiety Scale (HAM-A) Total Score
Description: The HAM-A is an anxiety rating scale consisting of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behavior at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total scores range from 0 to 56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe. Total scores above 30 are rare, but indicate very severe anxiety. Final Visit includes data from Week 52 or earlier for participants who didn't complete the 52 weeks.
Time Frame: Baseline and Weeks 4, 24 and 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Vortioxetine
Number analyzed (Participants) | 818
scores on a scale
  Week 4 (n=818) | -2.9 (5.12)
  Week 24 (n=642) | -5.1 (6.44)
  Week 52 (n=527) | -6.6 (6.38)
  Final Visit (n= 818) | -5.2 (6.76)

9. Secondary Outcome: Change From Baseline in the Clinical Global Impression of Severity of Illness Scale
Description: The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Considering total clinical experience, a patient is assessed on severity of mental illness on the following scale: 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill. Final Visit includes data from Week 52 or earlier for participants who didn't complete the 52 weeks.
Time Frame: Baseline and Weeks 4, 24 and 52
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Vortioxetine
Number analyzed (Participants) | 818
scores on a scale
  Week 4 (n=818) | -0.53 (1.002)
  Week 24 (n=642) | -0.98 (1.295)
  Week 52 (n= 527) | -1.33 (1.266)
  Final Visit (n=818) | -1.00 (1.338)

10. Secondary Outcome: Change From Baseline to the Final Visit in 36-item Short-form Health Survey (SF-36)
Description: The Medical Outcomes Study SF-36 is a participant self-rated questionnaire that is a general measure of perceived health status comprising 36 questions, which yields an 8-scale health profile. The 8 health concepts are: 1. Limitation in physical activities because of health problems. 2. Limitations in usual role activities because of physical health problems. 3. Bodily pain. 4. Limitations in social activities because of physical or emotional problems. 5. General mental health (psychological distress and well-being). 6. Limitations in usual role activities because of emotional problems. 7. Vitality (energy and fatigue). 8. General health perception. Each scale ranges from 0 (best) - 100 (worst).
Time Frame: Baseline and Week 52
Population: Participants in the safety analysis set who had at least 1 post-baseline efficacy measurement, and with available Final Visit data.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Vortioxetine
Number analyzed (Participants) | 824
scores on a scale
  Physical functioning subscore (n=824) | 4.5 (15.88)
  Role-physical subscore (n=824) | 8.1 (25.51)
  Bodily pain subscore (n=824) | 4.9 (24.29)
  General health subscore (n=823) | 6.4 (18.38)
  Vitality subscore (n=824) | 10.1 (23.03)
  Social functioning subscore (n=824) | 10.9 (26.90)
  Role-emotional subscore (n=824) | 12.3 (28.24)
  Mental health subscore (n=824) | 10.7 (22.04)

11. Secondary Outcome: Change From Baseline to the Final Visit in the Sheehan Disability Scale
Description: The Sheehan Disability Scale (SDS) assesses functional impairment in 3 domains: work/school, social life or leisure activities, and home life or family responsibilities. The participant rates the extent to which each aspect is impaired on a 10-point visual analog scale, from 0 (not at all) to 10 (extremely). The 3 scores are added together to calculate the total score, which ranges from 0 to 30, with higher scores indicating more impairment.
Time Frame: Baseline and Week 52
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Vortioxetine
Number analyzed (Participants) | 536
scores on a scale | -4.6 (8.01)

12. Secondary Outcome: Health Care Resource Utilization Assessed by the Health Economic Assessment Questionnaire
Description: Healthcare resource utilization was assessed by the Health Economic Assessment (HEA) questionnaire, which monitors participants absenteeism from work, as well as resource use such as visits to a general practitioner, outpatient and inpatient services, hospitalization, medications, and other relevant services over the past 8 weeks.
Time Frame: Baseline and Week 52
Population: Safety set with available data
Measure: Number; unit: participants
Arm/Group | Vortioxetine
Number analyzed (Participants) | 834
participants
  Baseline: Any resource use | 137
  Baseline: Any hospitalization-related services | 4
  Baseline: Hospitalization related to depression | 0
  Baseline: Any sick leave | 53
  Baseline: Sick leave related to depression | 42
  Week 52: Any resource use | 138
  Week 52:Any hospitalization-related services | 7
  Final Visit: Hospitalization related to depression | 0
  Week 52: Any sick leave | 41
  Week 52: Sick leave related to depression | 25

ADVERSE EVENTS:
Time Frame: From first dose of study until 30 days after the last dose.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Vortioxetine
Serious Adverse Events (participants affected / at risk) | 29/834
Other Adverse Events (participants affected / at risk) | 452/834
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vortioxetine (N=834)
Anemia (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Tachycardia paroxysmal (Cardiac disorders) | 1
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Edema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Abscess limb (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Influenza (Infections and infestations) | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Ischemic stroke (Nervous system disorders) | 1
Alcohol abuse (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Major depression (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 2
Abortion induced (Surgical and medical procedures) | 1
Uterine hemorrhage (Reproductive system and breast disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vortioxetine (N=834)
Nausea (Gastrointestinal disorders) | 127
Diarrhoea (Gastrointestinal disorders) | 60
Dry mouth (Gastrointestinal disorders) | 30
Dyspepsia (Gastrointestinal disorders) | 28
Constipation (Gastrointestinal disorders) | 25
Vomiting (Gastrointestinal disorders) | 25
Fatigue (General disorders) | 30
Nasopharyngitis (Infections and infestations) | 82
Upper respiratory tract infection (Infections and infestations) | 53
Influenza (Infections and infestations) | 33
Urinary tract infection (Infections and infestations) | 23
Bronchitis (Infections and infestations) | 19
Weight increased (Investigations) | 36
Back pain (Musculoskeletal and connective tissue disorders) | 32
Headache (Nervous system disorders) | 102
Dizziness (Nervous system disorders) | 57
Somnolence (Nervous system disorders) | 33
Insomnia (Psychiatric disorders) | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 17
Hypertension (Vascular disorders) | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.